CLINICAL TRIAL: NCT03644394
Title: Implantable MyoElectric Sensors (IMES) for Prosthetic Control in Transhumeral Amputees
Acronym: TH-IMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Salminger, Subinvestigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1320/2014
Record Dates: First submitted 2018-08-11; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Implantation (Other): Surgical Implantation of IMES sensors
  Interventions: Device: Implantation of IMES sensors

INTERVENTIONS:
Device: Implantation of IMES sensors — Surgical implantation of IMES sensors during routine surgery to improve prosthetic control

SUMMARY:
The Implantable Myoelectric Sensors (IMES) system is an investigational device intended to improve signal quality and consistency of myoelectric signals for prosthetic control in individuals suffering from an above elbow (transhumeral) amputation. The sensors pick up myoelectric signals intramuscularly and therefore signal quality is not affected from electrode replacement, perspiration, or artefacts.

DETAILED DESCRIPTION:
Implantable Myoelectric Sensors (IMES), the surgical tools implantation, and the external equipment used to control an electromechanical prosthetic device, together comprise the IMES System (investigational product, medical device).

Each IMES acts as an independent differential amplifier consisting of custom electronics housed within a biocompatible, hermetically sealed ceramic cylinder with metal end caps. The end caps serve as electrodes for picking up EMG activity during muscle contraction. Reverse telemetry (via a coil around the arm) is used to transfer data from the implanted sensor, and forward telemetry is used to transmit power and configuration settings to the sensors. The coil and associated electronics are housed within the frame of a prosthesis. A control system that sends data associated with muscle contraction to the motors of the prosthetic joints is housed in a belt-worn, battery-powered device. A cable attaches the control unit to the prosthetic frame.

An IMES is implanted into each targeted muscle that will be used to control a function of the prosthetic arm. Two IMES devices are needed for each DOF. For example, one device would control fingers opening and another device would control fingers closing.

ELIGIBILITY:
Inclusion Criteria:

* unilateral transhumeral amputation
* can speak and comprehend German
* undergone amputee rehabilitation, including being trained to wear and use a conventional myoelectric prosthesis
* residual upper limb meets the criterions for TMR surgery

Exclusion Criteria:

* Known genetic neuromuscular disorder
* bleeding or clotting disorder
* active implant
* any metal fragments or metal implants located within the residual upper limb stump
* Female patients if pregnant or breast-feeding

Ages: 16 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in hand function over time | at 3, 6, 9 and 12 months after final prosthetic fitting
  Southampton Hand Assessment Procedure

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hofer, PhD, Study Chair — Otto Bock

IPD SHARING:
Plan to Share IPD: No
The study including all results is already submitted to be published